CLINICAL TRIAL: NCT06951295
Title: Comparative Study Between Transcutaneous Ultrasonography and Direct Laryngoscopy for Assessment of Vocal Cord Mobility at the End of Thyroidectomy Operation
Acronym: Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MS 12/2023/2024
Record Dates: First submitted 2025-02-21; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Assessment of Vocal Cord Mobility; Thyroidectomy
Keywords: Thyroidectomy; Assessment of vocal cord mobility; Transcutanous ultrasonography
MeSH Terms: interventions — Thyroidectomy

STUDY DESIGN:
Intervention Model Description: At the same time of extubation investigator document the results and anesthesiologist record the results , they totally blind to results
Who Masked: Care Provider, Investigator
Masking Description: Investigator and anesthesiologist were blinded to results in the end of surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct laryngoscopy (Active Comparator): Direct laryngoscopy is a gold standard device to visualise the larynx and vocal cord mobility after thyroidectomy operation , that allows assessment of vocal cords mobility before extubation after thyroidectomy operation,we assess mobility with endotracheal tube and without endotracheal tube
  Interventions: Procedure: Thyroidectomy operation is a surgical removal of thyroid, injury of recurrent laryngeal nerve one of common complications of thyroidectomy Which can affect Vocal cords mobility
- Transcutanous ultrasonography (Active Comparator): Transcutanous ultrasonography is a tool non invasive reliable diagnostic method to assess vocal cords mobility , which can assess vocal cords mobility before extubation , that may be helpful to exclude recurrent laryngeal nerve injury as early as possible ,that may protect the patient from any possible complications
  Interventions: Procedure: Thyroidectomy operation is a surgical removal of thyroid, injury of recurrent laryngeal nerve one of common complications of thyroidectomy Which can affect Vocal cords mobility

INTERVENTIONS:
Procedure: Thyroidectomy operation is a surgical removal of thyroid, injury of recurrent laryngeal nerve one of common complications of thyroidectomy Which can affect Vocal cords mobility — Assessment of vocal cords mobility at thyroidectomy operation is very important and life saving for patient, during thyroidectomy one of common complications, injury of recurrent laryngeal nerve unilateral or bilateral, unilateral injury may complicate to dysphonia, bilateral injury may complicate to dyspnea
  Other Names: Thyroidectomy; Assessment of vocal cords mobility; Recurrent laryngeal nerve injury; Thyroidectomy operation

SUMMARY:
The aim of work of this study is to evaluate Transcutanous Ultrasonogrphy for assessment of vocal cord mobility in comparison to Direct laryngoscopy during extubation after thyroidectomy

DETAILED DESCRIPTION:
The aim of work of this study is to evaluate Transcutanous Ultrasonogrphy for assessment of vocal cord mobility in comparison to Direct laryngoscopy during extubation after thyroidectomyA. Preoperative settings: All patients will be assessed preoperatively by careful history taking, full physical examination, and laboratory evaluation and vocal cord mobility and voice quality be assessed by ENT and anesthesiologist by ultrasound.

B. Intraoperative settings:

On arrival of the patients to the operative room, electrocardiography, non-invasive blood pressure, and pulse oximetry will be applied. Baseline parameters such as heart rate (HR) , blood pressure (BP), and oxygen saturation (SpO2) will be also recorded.

Intravenous (IV) line will be inserted and IV lactated Ringer 500ml bolus then started as calculated by fluid chart. For both groups, General anesthesia will be performed After 3 minutes of pre- oxygenation, anaesthesia will be induced with IV 1 mcg/kg of fentanyl, 2 mg/kg of propofol and 0.5 mg/kg of atracurium to facilitate endotracheal intubation.

- Anesthesia will be maintained with 50% of oxygen in air, 1-2 % isoflurane and 0.1mg/kg atracurium every 20 minutes.

Both groups will receive rescue dose of fentanyl 0.5 mcg/kg for an increase in HR or MAP 20% above the baseline value. - All patients will be given IV 1 mg of granisetron and 40 mg of pantoprazole.

After end of surgery:

- Residual paralysis will be reversed with 0.05 mg/kg neostigmine and 0.02 mg/kg atropine. All patients underwent to two procedure mentioned above by two anesthesiologist.

Transcutanous ultrasonography by the investigator. Direct laryngeoscopy by the anesthesiologist. Transcutanous laryngeal ultrasonography: (TLUS) by using ultrasonogrphy sonosite 5- 10-MHz linear probe , patient 's position is supine with neck hyperextended in same position of surgery.Apply aseptic gel and sterile gloves to put probe on sutures .Probe is placed transversally on top of the thyroid cartilage to evaluate the vocal cords mobility.And move craniocaudal until two vocal cords are seen if difficult to find put probe on lateral side .True and false vocal cords will be seen, true will be hypoechoic below thyroid cartilage and false will be hyperechoic.When both true vocal cords move medially towards midline, this means NO nerve palsy.but when either one or both vocal cords not moved, this means there is nerve palsy. Direct Laryngeoscopy: Inserted in oral cavity and show both vocal cords mobility, if both mobile there is NO palsy , if one immobile and another mobile may be chance of stridor and if both immobile there is risk of airway obstruction. All results will be documented at the same time and comparison will be matched between the investigetor and the anesthesiologist and Statistical analysis will be done.

Postoperative settings: - All patients will continue to be monitored in the post- anesthesia care unit (PACU) for their HR normal range(60-100bpm), MAP normal(120/80)and SpO2> 95% on room air.

Analysis of voice change should be done by ability to speak and if there is any respiratory distress and by ENT consultation

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes patients aged above 21 years
2. BMI<40kg/m2
3. American Society of Anesthesiologists(ASA) Physical Status Class- II and class- III
4. Scheduled for elective thyroid surgery with intact vocal cords
5. Approved to give informed consent and preoperative assessment by ENT specialist using Indirect laryngoscopy.

Exclusion Criteria:

1. Patient refused to participate.
2. Morbid obesity (BMI: >40kg/m^2)
3. Age below 21 years.
4. American Society of Anesthesiologists(ASA) Physical Status Class IV.
5. Previous operation in thyroid gland.
6. Any previous vocal cords paralysis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Early assessment of vocal cord injury | Immediately after the surgery
  Early detection of any recurrant laryngeal nerve injury or paralysis at the end of surgery by vocal cords mobility examined by investigator by TLUS and by direct laryngeoscopy by anesthesiologist.

SECONDARY OUTCOMES:
Direct laryngoscopy adverse effects | Perioperatively
  more reliable and less adverse effects of transcutanous laryngeal ultrasonography.
Transcutanous laryngeal ultrasonography | Perioperatively
  Transcutanous laryngeal ultrasonography is comparable with direct laryngoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code